CLINICAL TRIAL: NCT07122310
Title: A Prospective, Randomized, Comparative Study of a 1064-nm Fractional Picosecond Laser Versus Intense Pulsed Light in Facial Rejuvenation
Brief Title: Comparative Study of a 1064-nm Fractional Picosecond Laser Versus IPL in Facial Rejuvenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Yanjun Dan, Resident Physician, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2022-824
Record Dates: First submitted 2025-08-05; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Skin Aging; Skin Rejuvenation; Photoaging
Keywords: Skin Rejuvenation; Picosecond laser; Intense pulsed light
MeSH Terms: interventions — Intense Pulsed Light Therapy

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned in a 1:1 ratio to receive either a 1064-nm fractional picosecond laser treatment or an intense pulsed light (IPL) treatment. Each group received three treatment sessions at 4-6 week intervals.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Picosecond Laser Group (Experimental)
  Interventions: Device: 1064-nm Fractional Picosecond Laser (PicoWay)
- Intense Pulsed Light (IPL) Group (Experimental)
  Interventions: Device: Intense Pulsed Light Therapy (M22 IPL System)

INTERVENTIONS:
Device: 1064-nm Fractional Picosecond Laser (PicoWay) — Intervention Name: 1064-nm Fractional Picosecond Laser (PicoWay) Participants in this group received full-face treatments using a PicoWay® laser system (Candela, Wayland, MA, USA) equipped with a 1064-nm RESOLVE fractional handpiece. Treatment parameters included a 6 mm spot size, 6 Hz repetition rate, 450 ps pulse duration, and energy settings ranging from 1.5 to 2.3 mJ per microbeam. Each session consisted of 2-3 passes (approximately 2000-4000 pulses), adjusted based on individual response. Three sessions were delivered at 4-6-week intervals. Cold compresses were applied for 20 minutes immediately post-treatment.
  Arms: Picosecond Laser Group
Device: Intense Pulsed Light Therapy (M22 IPL System) — Intervention Name: Intense Pulsed Light Therapy (M22 IPL System)
  Intervention Description:
  Participants in this group underwent full-face treatments using an M22® IPL system (Lumenis, Yokneam, Israel) with a 560 nm cutoff filter. Treatment parameters included a pulse duration of 3.5-4 ms, pulse delay of 25-30 ms, and fluence of 12-18 J/cm², adjusted based on individual response. Each treatment involved approximately 40-60 pulses. Three sessions were performed at 4-6-week intervals. A layer of medical ultrasound gel was applied before treatment and maintained for 15-20 minutes post-treatment.
  Arms: Intense Pulsed Light (IPL) Group

SUMMARY:
This is a single-center, prospective, randomized controlled trial conducted at Huashan Hospital, Fudan University. The purpose of this study is to compare the effectiveness and safety of two non-invasive treatment options-1064-nm fractional picosecond laser and intense pulsed light (IPL)-for facial rejuvenation. A total of 38 participants seeking cosmetic improvement were randomly assigned to receive three sessions of either picosecond laser or IPL treatment at 4-6 week intervals.

Each participant was monitored throughout the treatment period and at one month after the final session. The study assessed improvements in skin texture, pigmentation, and wrinkles, as well as treatment-related side effects. All participants provided informed consent and received standardized post-treatment care instructions, including moisturization and sun protection. The results of this study may help guide non-surgical treatment options for skin aging.

ELIGIBILITY:
Inclusion Criteria:

（1）Individuals aged 30-60 years with a GSP score of 1-4;（2）Fitzpatrick skin phototypes III-IV;（3）Written informed consent obtained.

Exclusion Criteria:

（1）Pregnant or lactating women;（2）Patients with severe systemic diseases;（3）Individuals with coagulation dysfunction;（4）Patients with mental disorders;（5）Photosensitive individuals;（6）Individuals with infections at the treatment site;（7）Individuals who have used photosensitive drugs within 4 weeks;（8）Individuals who have received other cosmetic treatments such as laser, intense pulsed light (IPL), radiofrequency, chemical peels (e.g., glycolic acid), fillers, etc., within 6 months;（9）Individuals with a personal or family history of keloids;（10）Individuals with a personal or family history of cutaneous squamous cell carcinoma or melanoma;（11）Individuals with a personal or family history of vitiligo;（12）Individuals with a history of intense sun exposure or ultraviolet (UV) radiation within 1 month.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2021-09-26 (Actual); Primary Completion 2023-01-08 (Actual); Study Completion 2023-06-19 (Actual)

PRIMARY OUTCOMES:
Blinded GSP (Global Score for Photoaging) assessment by two dermatologists | 1 month after third treatment (approximately 12-16 weeks after baseline)
  Global skin photoaging score assessed by blinded dermatologists using the Global Skin Photoaging (GSP) Scale. Scale range: 0-4, where higher scores indicate more severe photoaging.

SECONDARY OUTCOMES:
Blinded GSP scoring | baseline (before first treatment), before second treatment (approximately 4-6 weeks after baseline), before third treatment (approximately 8-12 weeks after baseline)
  Global skin photoaging score assessed by blinded dermatologists using the Global Skin Photoaging (GSP) Scale. Scale range: 0-4, where higher scores indicate more severe photoaging.
  The scoring criteria are defined as follows:
  0: Smooth skin without visible wrinkles or pigmentary heterogeneity in cheeks, forehead, or perioral regions
  1. Discrete focus of textural roughness, dyschromia, or fine lines in one facial region (cheeks/forehead/perioral)
  2. Two distinct areas demonstrating textural roughness, dyschromia, or fine lines; OR concurrent manifestations (roughness + dyschromia + wrinkles) in one region
  3. Three affected areas; OR concurrent manifestations in two regions
  4. Photodamage exceeding grade 3 criteria
Regional Fine Line and Dyschromia Grading by Dermatologists | before second treatment (approximately 4-6 weeks after baseline), before third treatment (approximately 8-12 weeks after baseline), and 1 month after third treatment (approximately 12-16 weeks after baseline)
  Fine lines graded on the Modified Fine Line Improvement Scale (-1 to 4: -1=worsening, 0=no change, 1=1-25% improvement, 2=25-50%, 3=50-75%, 4=75-100%; higher scores = greater improvement).
  Dyschromia graded on the Modified Dyschromia Improvement Scale (-1 to 4: -1=increased severity, 0=no change, 1=1-25% reduction, 2=25-50% reduction, 3=50-75% reduction, 4=75-99% reduction; higher scores = greater improvement).
Quantitative Assessment of Skin Roughness Using C-Cube Imaging System | baseline (before first treatment), before second treatment (~4-6 weeks after baseline), before third treatment (~8-12 weeks), and 1 month after third treatment (~12-16 weeks)
  Skin surface roughness will be objectively quantified using the C-Cube high-resolution imaging system (Pixience, Toulouse, France). Standardized images will be captured from predefined facial regions (e.g., cheek or forehead) under consistent lighting and positioning conditions. Roughness values will be automatically calculated by the system's built-in analysis software. Measurements will be performed at baseline, second, third, and fourth follow-up visits to monitor treatment-induced changes.
Quantitative Skin Pigmentation and Erythema Assessment Using SkinColorCatch | baseline (before first treatment), before second treatment (~4-6 weeks after baseline), before third treatment (~8-12 weeks), and 1 month after third treatment (~12-16 weeks)
  Objective colorimetric measurements will be performed using the Delfin SkinColorCatch® device to quantify skin pigmentation and erythema in predefined facial regions. The following parameters will be recorded at each time point: Melanin Index (MI), L* value (lightness), and Erythema Index (EI). Measurements will be obtained under standardized ambient lighting and positioning conditions at baseline, second, third, and fourth follow-up visits.
Transepidermal Water Loss (TEWL) Measurement Using Delfin Vapometer | baseline (before first treatment), before second treatment (~4-6 weeks after baseline), before third treatment (~8-12 weeks), and 1 month after third treatment (~12-16 weeks)
  Skin barrier function will be assessed by measuring transepidermal water loss (TEWL) using the Delfin Vapometer® device. Measurements will be taken at standardized facial sites under controlled environmental conditions (temperature and humidity) following device guidelines. TEWL values will be recorded at baseline and at the second, third, and fourth follow-up visits to evaluate changes in skin barrier integrity over the treatment course.
Standardized VISIA Photographic Documentation | baseline (before first treatment), before second treatment (~4-6 weeks after baseline), before third treatment (~8-12 weeks), and 1 month after third treatment (~12-16 weeks)
  Standardized facial photographs will be captured using the VISIA Complexion Analysis System (Canfield Scientific, USA) at each time point to document changes in skin appearance. The system will provide consistent image capture under controlled lighting and positioning conditions. VISIA documentation will support visual assessment of treatment-related changes in texture, pores, pigmentation, and overall skin condition. Images will be used for qualitative reference and supplemental analysis by blinded evaluators.
Incidence of Adverse Events | before second treatment (~4-6 weeks after baseline), before third treatment (~8-12 weeks), and 1 month after third treatment (~12-16 weeks)
  Adverse events (AEs) including erythema, edema, hyperpigmentation, hypopigmentation, burning sensation, pain, and scarring will be recorded following each treatment session and at each follow-up visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this single-center study does not have a formal data sharing infrastructure, and participants did not provide consent for public data sharing. Aggregated results may be reported in publications or upon reasonable request.

REFERENCES:
- [Derived] Zhang J, Wu C, Liu Y, Yan F, Chen Q, Zhu Y, Xiang LF, Ren J. Comparative Study of a 1064 nm Fractional Picosecond Laser Versus Intense Pulsed Light in Facial Rejuvenation: A Prospective Randomized Trial. Lasers Surg Med. 2026 Jan 4. doi: 10.1002/lsm.70094. Online ahead of print. PMID 41485124